CLINICAL TRIAL: NCT00065871
Title: Improving Contraceptive Practice and Delivery Through Community Pharmacists: The Direct Access Study
Brief Title: The Direct Access Study: Access to Hormonal Birth Control Through Community Pharmacies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Prevention
Other Study IDs: HD42427
Record Dates: First submitted 2003-08-01; First posted 2003-08-05 (Estimated); Last update posted 2007-04-06 (Estimated); Status verified 2004-11

CONDITIONS: Contraception
Keywords: Pharmacist prescribers; Increased access; Hormonal contraception; Birth control pills; Birth control patch; Vaginal contraceptive ring

INTERVENTIONS:
Behavioral: Contraceptive Screening by Pharmacist
Behavioral: Contraceptive Prescribing by Pharmacist

SUMMARY:
Hormonal birth control methods include birth control pills, patches, and vaginal rings; they are normally available only with a doctor's prescription. This study will evaluate a program designed to increase the availability of birth control by allowing pharmacists to give women hormonal birth control without a doctor's prescription. Under this program, pharmacists will evaluate women who want to use birth control according to specific guidelines created by doctors. If a woman meets the criteria in the guidelines, a pharmacist could then give her the appropriate form of hormonal birth control.

DETAILED DESCRIPTION:
The Institute of Medicine's Committee on Unintended Pregnancy urges increasing access to contraception through broadening the range of health professionals that provide birth control. Evidence-based family planning practice no longer requires a physical examination before prescribing hormonal contraceptives to women. Community pharmacists efficiently provide emergency contraceptive pills (ECP) and women report satisfaction with the direct access. These women, as well as many women purchasing less effective over-the-counter (OTC) contraceptive methods, could benefit from more pharmacist-dispensed birth control choices, such as hormonal methods. The Direct Access Study will assess the feasibility of pharmacists, under Collaborative Drug Therapy Agreements with independent prescribers, providing hormonal contraceptives in community pharmacies. Specifically, the study will evaluate the impact upon hormonal contraception initiation and continuation rates when women's care is managed by pharmacists.

Using Collaborative Drug Therapy Agreements jointly developed with licensed prescribers (physicians and nurse practitioners), pharmacists in four Fred Meyer pharmacies will identify women who are at risk of unintended pregnancy and will offer to evaluate them for their suitability to safely use oral contraceptives, contraceptive patches, or the contraceptive vaginal ring. Through self-administered medical and contraceptive history questionnaires, interested women will select the most suitable contraceptive methods. Pharmacists will then complete the screening process and prescribe hormonal contraceptives according to the protocol guidelines.

Pharmacists will encourage women to follow up with a primary care practitioner or family planning clinic for cervical exams and reproductive tract infection screening as indicated. Pharmacists will have authority to provide an initial 3-month prescription and an additional 9-month prescription if blood pressure is normal at a three-month revisit. Effectiveness of pharmacists' interventions will be measured by initiation and continuation of hormonal methods by women to whom pharmacists have offered them. Feasibility will be determined by measurement of both acceptability and sustainability. Acceptability will be measured by surveys of women, pharmacists, and prescribers. Sustainability will be measured by economic and work-flow outcomes for the pharmacies, including evidence that women, private third-party payers, and public payers are willing to pay for the services. If safety is documented after preliminary analysis, injectable contraceptive methods will be added to the study.

ELIGIBILITY:
Inclusion Criteria

* At risk for unintended pregnancy
* Access to participating Fred Meyer Pharmacy
* English-speaking
* Health insurance or ability to pay for contraceptive care

Exclusion Criteria

* Age less than 18 years
* Age greater than 45 years
* Unable to become pregnant
* Not English speaking
* Not planning to remain in area
* Not planning to use the same pharmacy
* Unable to pay for services

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250
Dates: Start 2003-06; Study Completion 2006-02

PRIMARY OUTCOMES:
The number and characteristics of women who seek hormonal contraceptives from pharmacists as evidenced by study consent or enrollment.
The number and characteristics of women not able to obtain hormonal contraceptives due to contraindications, costs, etc.
The proportion and characteristics of those women who continue to use the initial method after 3, 6, and 12-months compared with national literature and with women who do not obtain the method by direct pharmacist access.
Safety evaluation to include prescribing protocol adherence (no women with absolute contraindication given estrogen; blood pressure monitoring done prior to more than three cycles of estrogen methods; no woman given a hormonal method while pregnant.

SECONDARY OUTCOMES:
The number and characteristics of women who choose hormonal contraceptives for the first time compared to national literature.
The amount of time required for pharmacists to be trained and to conduct the defined interventions in the course of their ongoing pharmach practice.
The number and characteristics of eligible Medicaid waiver applicants enrolled by pharmacists compared with state figures for other providers.
The proportion of billed insurance claims that are paid.
The number and types of referrals to clinicians made by pharmacists and the proportion of counseled clients who follow through on the referrals that were made.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Gardner, PhD, Principal Investigator — University of Washington
Locations (5):
- United States (5):
  - Fred Meyer Pharmacy, Kent, Washington
  - Fred Meyer Pharmacy, Kirkland, Washington
  - Fred Meyer Pharmacy, Puyallup-South Hill, Washington
  - Bartell Drugs, University Village, Seattle, Washington
  - Fred Meyer Pharmacy, Seattle-Broadway, Washington

REFERENCES:
- [Background] Stewart FH, Harper CC, Ellertson CE, Grimes DA, Sawaya GF, Trussell J. Clinical breast and pelvic examination requirements for hormonal contraception: Current practice vs evidence. JAMA. 2001 May 2;285(17):2232-9. doi: 10.1001/jama.285.17.2232. PMID 11325325
- [Background] Gardner JS, Hutchings J, Fuller TS, Downing D. Increasing access to emergency contraception through community pharmacies: lessons from Washington State. Fam Plann Perspect. 2001 Jul-Aug;33(4):172-5. No abstract available. PMID 11496935
- [Background] Faculty of Family Planning and Reproductive Health Care. Royal College of Obstetricians and Gynaecologists. First prescription of combined oral contraception: recommendations for clinical practice. Br J Fam Plann. 2000 Jan;26(1):27-38. No abstract available. PMID 10819591